CLINICAL TRIAL: NCT02210312
Title: Are Preoperative Depressive Symptoms Predictive for Postoperative Dysfunction in Non-cardiac Surgery?
Brief Title: Study of Depressive Symptoms Predicting Postoperative Cognitive Dysfunction
Acronym: DeprPOCD
Status: Completed | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Other Study IDs: PV4646
Record Dates: First submitted 2014-06-16; First posted 2014-08-06 (Estimated); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium; Depressive Symptoms
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- elective non-cardiac surgery and non-neurosurgical procedures: 300 Patients aged 60 years and older undergoing elective non-cardiac surgery and non-neurosurgical procedures in general anaesthesia or combined general/regional anaesthesia with a duration of operation of 120 minutes or longer. 80 age-, gender- and education-matched healthy controls.

SUMMARY:
Postoperative cognitive dysfunction (POCD) describes a condition where cognitive functions such as attention, perception, concentration, learning, abstract thinking and problem solving are impaired postoperatively. These changes can be resolved after weeks and months. In some cases, changes are permanent.

DETAILED DESCRIPTION:
The aetiology of POCD is multifactorial. One described risk factor is preoperative existing depressive symptoms in patients undergoing cardiac surgery.

A total of 300 consecutive patients and 80 healthy controls will be enrolled in this study. Patients will be followed up at 7 days, 3 months and 1 year postoperatively. The co gnitive function will be tested and compared to tests done before surgery. Postoperatively - from the day of operation until the 7th day (except day 6) - grade of sedation, agitation, signs of delirium, pain, cardiac, respiratory, renal and infectious complications will be monitored.

Next to preoperative depressive symptoms we will also evaluate a diagnosed depression, anxiety, pain, health-related quality of life, physical comorbidities, adrenal cortical insufficiency, type of anaesthesia, intraoperative blood loss, organ complications, postoperative delirium, baseline cognitive functioning and the number of operations/anaesthetics in the study period after the initial operation as further potential predictors of POCD.

In addition, laboratory values and certain medications will be documented. These include: anaemia, hypercalcaemia, thyroidal gland hormones, electrolytes, creatinine, urea, glomerular filtration rate and cortisone therapy.

ELIGIBILITY:
Inclusion Criteria for patients and healthy controls:

* Age > 60 years
* Written informed patient's consent

Additional Inclusion Criteria for patients:

* Elective non-cardiac surgery and non-neurosurgical procedures in general anaesthesia or combined general/regional anaesthesia
* Minimum of duration of operation 120 minutes
* Baseline testing 3-14 days preoperatively

Additional Inclusion Criteria for healthy controls:

* matched for age, gender and education
* no surgery over the study period

Exclusion Criteria for patients and healthy control:

* German not mother tongue
* Illiteracy
* Mental disability
* Vision impairment not correctable
* Hearing impairment not correctable
* Illegal substance abuse (current or past history)
* Alcohol abuse (current or past history)
* Chronic benzodiazepine use
* Psychosis (current or past history)
* Parkinson Disease
* Dementia
* Multiple sclerosis
* Epilepsy (current or past history)
* Cerebral tumor (current or past history)
* Apoplexy or intracranial bleeding (current or past history)
* Severe traumatic brain injury (current or past history)
* Severe liver disease (Child Pugh B, C, liver insufficiency)
* Severe kidney disease with dialysis
* Mini Mental Status Examination < 24 points

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female and male patients, aged 60 years and older undergoing elective non-cardiac surgery and non-neurosurgical procedures in general anaesthesia or combined general/regional anaesthesia. To correct for practice effects and conduct additional comparisons, 80 healthy controls will be enrolled and assessed at the same time points (neuropsychological tests and questionnaires).
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-05; Primary Completion 2018-07 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Frequency of occurrence of early POCD | 7 days
  POCD is measured by use of a neuropsychological test battery comprising the following subtests: Alertness, Go/Nogo, and Incompatibility from the TAP 2.3 (attention), Trail Making Test A and B (attention), Digit span (memory), Verbal Learning and Memory Test (memory), Regensburg Word Fluency Test (executive function)
Frequency of occurrence of intermediate POCD | 3 months
  POCD is measured by use of a neuropsychological test battery comprising the following subtests: Alertness, Go/Nogo, and Incompatibility from the TAP 2.3 (attention), Trail Making Test A and B (attention), Digit span (memory), Verbal Learning and Memory Test (memory), Regensburg Word Fluency Test (executive function)
Frequency of occurrence of late POCD | 1 year
  POCD is measured by use of a neuropsychological test battery comprising the following subtests: Alertness, Go/Nogo, and Incompatibility from the TAP 2.3 (attention), Trail Making Test A and B (attention), Digit span (memory), Verbal Learning and Memory Test (memory), Regensburg Word Fluency Test (executive function)

SECONDARY OUTCOMES:
Frequency of occurrence of postoperative delirium | 7th postoperative day
  measured twice per day: Confusion Assessment Method (CAM-ICU) and Richmond Agitation and Sedation Scale (RASS)
Rate of organ complications (cardiac, respiratory, renal) | day of operation until 7th postoperative day
Hospital length of stay | day of admission until day of discharge, up to 24 weeks
Mortality | 1 year
Health related quality of life | 7 days, 3 months, 1 year after operation
  Time Frame: 7 days after operation [Measure: Short Form-12 Health Survey: Item General Health] Time Frame: 3 months after operation [Measure: Short Form-12 Health Survey: Physical and mental health summary measures] Time Frame: 1 year after operation [Measure: Short Form-12 Health Survey: Physical and mental health summary measures]

OTHER OUTCOMES:
Dementia | Change from baseline sum score on the Mini-Mental State Examination (2nd ed.) [Time Frame: Before operation to 7 days, 3 months and 1 year after operation].
Preoperative depressive symptoms and anxiety | Baseline
  Preoperative depressive symptoms and anxiety are assessed with the Hospital Anxiety and Depression Scale (HADS). The HADS comprises 14 Items and 2 subscales with 7 items each. The items are answered on a 4-point rating scale from 0 to 3 with a scale score varying between 0 and 21. Higher scores represent higher distress (cut-off- scores: 0-7 = normal, 8-10 = borderline, 11-14 = severe symptoms, >=15 = very severe symptoms).
Past or present diagnosed depression | Baseline
  A self-administered questionnaire was developed to explore pre-existing depression (current or in past medical history) and its medical or/and non-medical treatment.
Pre- and perioperative pain | Baseline and interval from day of operation to day 7 after operation
  Preoperative pain: Numerical Rating Scale from 0 to 10 [Time Frame: Baseline] Perioperative pain: Numerical Rating Scale from 0 to 10, averaged over one week [Time Frame: Interval from day of operation to day 7 after operation]
Premorbid Intelligence | Baseline
  Multiple-Choice Vocabulary Intelligence Test (MWT-B, sum score)
Preoperative cognitive functioning | Baseline
  Global mean z-score on the neuropsychological test battery
Postoperative depressive symptoms and anxiety | 7 days, 3 months
  HADS, depression scale score [Time Frame: 7 days and 3 months after operation] HADS, anxiety scale score [Time Frame: 7 days and 3 months after operation]
Change in depressive symptoms and anxiety from baseline to 1 year | Change from baseline scale scores on the HADS depression and anxiety subscales [Time Frame: Before operation to 7 days, 3 months and 1 year after operation].

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wiede, MD, Principal Investigator — Department of Anaesthesiology and Intensive Care Medicine, University Hospital Hamburg Eppendorf
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, University Hospital Hamburg Eppendorf, Univ.-Prof. Dr. med. Alwin E. Goetz and Prof. Dr. med. Christian Zoellner, Hamburg, Germany